CLINICAL TRIAL: NCT06586021
Title: SEAL - Safety & Feasibility Evaluation of the Aortoseal™ for Seal and Fixation of Abdominal Aortic Aneurysms (AAA) Endovascular Grafts to the Aortic Wall"
Brief Title: Evaluation of the Aortoseal™ for Sealing and Fixation of AAA Endovascular Grafts to Aortic Wall
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endoron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 305CLD
Record Dates: First submitted 2024-09-02; First posted 2024-09-19 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Aortic Aneurysm (AAA)
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Aortoseal Endostapling System (Experimental): Prospective, early feasibility, non-randomized, single arm, multi-center, open-label clinical study
  Interventions: Device: Aortoseal Endostapling System

INTERVENTIONS:
Device: Aortoseal Endostapling System — Aortoseal Endostapling System

SUMMARY:
The Aortoseal Endostapling System is indicated in patients undergoing, or having undergone, treatment of an abdominal aortic aneurysm (AAA) with an endovascular graft to provide enhanced fixation and apposition to the aorta.

DETAILED DESCRIPTION:
The device may be implanted at the time of the initial endovascular graft procedure to maintain, or during a secondary procedure to restore, adequate aneurysm.

The study includes 5 years of follow-up, with visits at 30 days, 6 months, 1 year, and yearly thereafter through 5-years.

Follow-up assessments: Physical examination, X-ray, CT (with and without contrast) and assessments of any adverse events.

ELIGIBILITY:
Subjects diagnosed with a qualifying AAA suitable for elective endovascular repair with Endovascular Graft System or have a previously placed endovascular graft.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Adverse Events | through 5 years
  The EFS does not have defined primary endpoints nor any powered endpoints. The SEAL Study is not hypothesis driven. All endpoints will be analyzed descriptively
Access Site Complications | through 30 days
  The EFS does not have defined primary endpoints nor any powered endpoints. The SEAL Study is not hypothesis driven. All endpoints will be analyzed descriptively
All Adverse Events | through 5 years
  The EFS does not have defined primary endpoints nor any powered endpoints. The SEAL Study is not hypothesis driven. All endpoints will be analyzed descriptively
Endpoints related to Aortoseal Endostapling System | through 5 years
  The EFS does not have defined primary endpoints nor any powered endpoints. The SEAL Study is not hypothesis driven. All endpoints will be analyzed descriptively
Device Technical Success | during procedure
  The EFS does not have defined primary endpoints nor any powered endpoints. The SEAL Study is not hypothesis driven. All endpoints will be analyzed descriptively

CONTACTS AND LOCATIONS:
Locations (1):
- Sentara Health Research Center, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No